CLINICAL TRIAL: NCT03315247
Title: Telephone-Based Cognitive Behavioural Therapy for Post-Operative Bariatric Surgery Patients: A Randomized Controlled Trial
Brief Title: Tele-CBT Following Bariatric Surgery: Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Sanjeev Sockalingam, Deputy Psychiatrist-in-Chief, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-5655; 376045 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2017-08-31; First posted 2017-10-20 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Obesity
Keywords: Obesity; Bariatric Surgery; Bariatrics; Cognitive Therapy; Binge Eating
MeSH Terms: conditions — Obesity; Bulimia

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (No Intervention): Participants assigned to the Treatment as Usual group will attend routine clinic visits at the Toronto Western Hospital Bariatrics Surgery Program (TWH-BSP). These visits generally include education on bariatric surgery and nutrition. Patients meet with select members of the multidisciplinary team at 1, 2, and 3 years post-surgery, and may attend an optional monthly support group. Participants' service utilization (i.e., attendance at optional sessions) will be documented and compared across groups.
- Telephone-Based CBT (Experimental): The Tele-CBT intervention will be delivered 1 year following bariatric surgery. Participants will receive 6 weekly Telephone-based Cognitive Behavioural Therapy sessions and 1 final "booster" session 1 month later, all approximately 55-minutes in duration and scheduled at a time convenient for the participants.
  Interventions: Behavioral: Telephone-Based CBT

INTERVENTIONS:
Behavioral: Telephone-Based CBT — The Tele-CBT sessions focus on introducing the cognitive behavioural model of overeating and obesity, scheduling healthy meals and snacks at regular time intervals and recording consumption using food records, scheduling pleasurable alternative activities to overeating, identifying and planning for difficult eating scenarios, and reducing vulnerability to overeating by solving problems and challenging negative thoughts. Participants are expected to complete CBT homework between sessions, such as completing food records, engaging in pleasurable and self-care activities, and completing a variety of worksheets.
  Other Names: Tele-CBT
  Arms: Telephone-Based CBT

SUMMARY:
Bariatric (weight loss) surgery is the most effective treatment for extreme obesity, but surgery does not treat underlying psychological and behavioural issues. Currently, psychotherapy ("talk therapy") for eating problems is not routinely offered with surgery, and many people start to regain weight one year later. Objective: This study will examine if adding a convenient and accessible psychotherapy by phone one year after surgery will lead to increased weight loss two years after surgery. Primary Hypothesis: Relative to the Control group (who will get routine care), the group of individuals who get psychotherapy will have lower weights 2 years after surgery. Secondary Hypotheses: Relative to the Control group, the psychotherapy group will report significantly less maladaptive eating behaviours and medical burden, and significantly greater quality of life. Method: Participants recruited from the Bariatric Surgery Programs at Toronto Western Hospital will be randomly assigned to 1 of 2 groups: 1) Control (Usual Standard of Care) or 2) Tele-CBT (a 7-session telephone-based cognitive behavioural therapy [a type of "talk therapy"] intervention focused on developing coping skills to improve maladaptive thoughts, emotions, and eating behaviours, specifically designed for bariatric surgery patients, delivered 1 year post-surgery). They will have their weight measured and will complete measures of eating behaviour and quality of life prior to the intervention, and again at several time points extending to 2 years post-surgery. Implications: If Telephone-Cognitive Behavioural Therapy (CBT) is found to improve bariatric surgery outcomes, it could become the standard of care in Canadian bariatric surgery programs and beyond, and be routinely offered to patients who cannot feasibly attend CBT sessions due to physical or practical barriers.

ELIGIBILITY:
Inclusion Criteria:

* Received bariatric surgery 1 year ago
* Fluent in English
* Have Internet access to complete online questionnaires.

Exclusion Criteria:

* Current active suicidal ideation
* Current poorly controlled psychiatric illness that would render Tele-CBT very difficult, including serious mental illness (i.e., psychotic disorder, bipolar disorder), severe depression (i.e., current major depressive episode diagnosis and Patient Health Questionnaire [PHQ-9]61 score > 20), or severe anxiety (i.e., current anxiety disorder diagnosis and Generalized Anxiety Disorder [GAD-7]62 score >15)
* Current poorly controlled medical illness that would render Tele-CBT very difficult.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Weight | 1.25, 1.5, 2, 3 years post-surgery
  Change in weight measured in kg

SECONDARY OUTCOMES:
Changes in obesity-related medical comorbidities - Medication Burden | 2 and 3 years post-surgery
  Medication pill burden/Type 2 Diabetes Mellitus (T2DM) specific medication burden
Changes in obesity-related medical comorbidities - Medical Treatments | 2 and 3 years post-surgery
  Discontinuation of medical treatments
Changes in obesity-related medical comorbidities - T2DM | 2 and 3 years post-surgery
  Remission of T2DM (normalization of lab values discontinuation of medical treatments and remission of T2DM/normalization of lab values)
Changes in eating pathology - Emotional Eating | 1.25, 1.5, 2, and 3 years post-surgery
  Measured by the Emotional Eating Scale (EES). The EES is a 25-item self-report measure that assesses the tendency to cope with negative affect by eating. Respondents are presented with 25 emotions and are asked to rate the strength of their urge to eat on a scale from 1 (no desire to eat) to 5 (an overwhelming urge to eat) when experiencing each of the emotions. The total EES score is calculated as a sum of all 25 self-report answers. The EES consists of 3 subscales reflecting anger/frustration, anxiety, and depression. The EES subscale scores are calculated as a sum of all self-report answers of emotions that fall within the subscale categories.
Changes in eating pathology - Binge Eating | 1.25, 1.5, 2, and 3 years post-surgery
  Measured by the Binge Eating Scale (BES). The BES is a 16-item self-report measure that assesses the presence of binge eating behaviour indicative of an eating disorder. It was devised specifically for use with obese individuals. Respondents are asked to rate the way they feel about their eating behaviour from 1 (statements indicating they see no problem with their eating behaviour) to 4 (statements indicating they see a severe problem with their eating behaviour). Scores on the BES range from 0 to 46 with the total score calculated as a sum of all 16 self-report answers. Moderate and severe levels of binge eating correspond to cut-off scores of 18 and 27.
Changes in eating pathology - Loss of Control | 1.25, 1.5, 2, and 3 years post-surgery
  Measured by the Loss of Control over Eating Scale (LOCES-Brief). The LOCES-Brief is a 7-item self-report measure that assesses the behavioural and cognitive aspects of loss of control eating, which may occur even in the absence of objectively large eating binges. Respondents are asked to rate the frequency with which they have experienced loss of control over eating over the last month on a scale ranging from 1 (never) to 5 (always). Scores on the LOCES-Brief can range from 7 to 35 with the total score calculated as a sum of all 7 self-report answers.
Changes in eating pathology - Depression | 1.25, 1.5, 2, and 3 years post-surgery
  Measured by the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a 9-item self-report measure of depression severity. Respondents are asked to rate the frequency with which they have experienced depressive symptoms over the last two weeks on a scale ranging from 0 (not at all) to 3 (nearly every day). Scores on the PHQ-9 can range from 0 to 27 with the total score calculated as a sum of all 9 self-report answers. Mild, moderate, moderately severe, and severe levels of depressive symptoms correspond to cut-off scores of 5, 10, 15, and 20 respectively.
Changes in eating pathology - Quality of Life | 1.25, 1.5, 2, and 3 years post-surgery
  Measured by the EuroQol (EQ-5D-5L). The EQ-5D-5L is a 25 item self-report measure of health-related quality of life. The EQ-5D-5L covers the 5 domains of mobility, self-care, daily activities, pain/discomfort, and anxiety/depression. Each domain consists of 5 statements ranging from "I have no problems" to "I am unable to/I have extreme problems". Respondents are also asked to rate how good or bad their health is at the current point in time on a scale from 0 (worst health you can imagine) to 100 (best health you can imagine).
Changes in eating pathology - Anxiety | 1.25, 1.5, 2, and 3 years post-surgery
  Measured by the Generalized Anxiety Disorder Scale (GAD-7). The GAD-7 is a 7-item self report measure of anxiety severity. It was originally developed to diagnose generalized anxiety disorder, but it has also proved to be a good screening instrument for other disorders including panic disorder, social phobia, and post-traumatic stress disorder. Respondents are asked to rate the frequency with which they have experienced anxiety symptoms over the last two weeks on a scale ranging from 0 (not at all) to 3 (nearly every day). Scores on the GAD-7 can range from 0 to 21 with the total score calculated as a sum of all 7 self-report answers. Mild, moderate, and severe levels of anxiety symptoms correspond to cut-off scores on 5, 10, and 15 respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Sockalingam, MD, FRCPC, Principal Investigator — University of Toronto, University Health Network; Stephanie Cassin, PhD, CPsych, Principal Investigator — Toronto Metropolitan University; Raed Hawa, MD, FRCPC, Study Director — University of Toronto, University Health Network; Susan Wnuk, PhD, CPsych, Study Director — University of Toronto, University Health Network; Timothy Jackson, MD, FRCPC, Study Director — University of Toronto, University Health Network; Lorraine Lipscombe, MD, FRCPC, Study Director — Women's College Hospital; Allan Okrainec, MD, FRCPC, Study Director — University of Toronto, University Health Network; George Tomlinson, PhD, Study Director — University of Toronto; David Urbach, MD, FRCPC, Study Director — University of Toronto, University Health Network
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly in order to protect patient confidentiality. Aggregate and anonymous data will be shared in peer reviewed journal articles and scientific presentations.

REFERENCES:
- [Background] Meany G, Conceicao E, Mitchell JE. Binge eating, binge eating disorder and loss of control eating: effects on weight outcomes after bariatric surgery. Eur Eat Disord Rev. 2014 Mar;22(2):87-91. doi: 10.1002/erv.2273. PMID 24347539
- [Background] Sheets CS, Peat CM, Berg KC, White EK, Bocchieri-Ricciardi L, Chen EY, Mitchell JE. Post-operative psychosocial predictors of outcome in bariatric surgery. Obes Surg. 2015 Feb;25(2):330-45. doi: 10.1007/s11695-014-1490-9. PMID 25381119
- [Background] DiGiorgi M, Rosen DJ, Choi JJ, Milone L, Schrope B, Olivero-Rivera L, Restuccia N, Yuen S, Fisk M, Inabnet WB, Bessler M. Re-emergence of diabetes after gastric bypass in patients with mid- to long-term follow-up. Surg Obes Relat Dis. 2010 May-Jun;6(3):249-53. doi: 10.1016/j.soard.2009.09.019. Epub 2009 Oct 29. PMID 20510288
- [Background] Shah M, Simha V, Garg A. Review: long-term impact of bariatric surgery on body weight, comorbidities, and nutritional status. J Clin Endocrinol Metab. 2006 Nov;91(11):4223-31. doi: 10.1210/jc.2006-0557. Epub 2006 Sep 5. PMID 16954156
- [Derived] Cassin SE, Park KE, Leung SE, Ma C, Tomlinson G, Hawa R, Wnuk S, Jackson T, Urbach D, Okrainec A, Brown J, Sandre D, Sockalingam S. A Randomized-Controlled Trial Examining Telephone-Based Cognitive Behavioral Therapy for Patients After Metabolic and Bariatric Surgery: 18 Month Follow-up Results. Obes Surg. 2025 Oct;35(10):4103-4113. doi: 10.1007/s11695-025-08163-2. Epub 2025 Sep 1. PMID 40887513
- [Derived] Sockalingam S, Leung SE, Ma C, Tomlinson G, Hawa R, Wnuk S, Jackson T, Urbach D, Okrainec A, Brown J, Sandre D, Cassin SE. Efficacy of Telephone-Based Cognitive Behavioral Therapy for Weight Loss, Disordered Eating, and Psychological Distress After Bariatric Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2327099. doi: 10.1001/jamanetworkopen.2023.27099. PMID 37535357
- [Derived] Sockalingam S, Leung SE, Ma C, Hawa R, Wnuk S, Dash S, Jackson T, Cassin SE. The Impact of Telephone-Based Cognitive Behavioral Therapy on Mental Health Distress and Disordered Eating Among Bariatric Surgery Patients During COVID-19: Preliminary Results from a Multisite Randomized Controlled Trial. Obes Surg. 2022 Jun;32(6):1884-1894. doi: 10.1007/s11695-022-05981-6. Epub 2022 Feb 25. PMID 35218006